CLINICAL TRIAL: NCT05268692
Title: Neoadjuvant Chemotherapy for Pancreatic Cancer; GS vs. GnP
Brief Title: Neoadjuvant Chemotherapy for Pancreatic Cancer Followed by GS and GnP
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Kochi University (Other)
Responsible Party: Principal Investigator, Takehiro Okabayashi, Department of Surgery, Kochi University
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GSGnP
Record Dates: First submitted 2022-02-01; First posted 2022-03-07 (Actual); Last update posted 2022-03-07 (Actual); Status verified 2022-02

CONDITIONS: Pancreatic Adenocarcinoma
Keywords: Neoadjuvant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- GS (Active Comparator): gemcitabine plus S-1
  Interventions: Drug: GS
- GnP (Active Comparator): gemcitabine plus nab-paclitaxel
  Interventions: Drug: GnP

INTERVENTIONS:
Drug: GS — drip infusion of gemcitabine plus oral administration of S-1 S-1 received S-1 orally twice daily at a dose calculated according to body-surface area (BSA) (< 1.25 m2, 60 mg/d; ≥ 1.25 to < 1.5 m2, 80 mg/d; ≥ 1.5 m2, 100 mg/d) on days 1 through 14 of a 21-day cycle gemcitabine received gemcitabine intravenously at a dose of 800 mg/m2 over 30 minutes on days 1 and 8of a 21-day cycle.
  Arms: GS
Drug: GnP — drip infusion of both gemcitabine and nab-paclitacel gemcitabine received gemcitabine intravenously at a dose of 800 mg/m2 over 30 minutes on days 1, 8, and 15 of a 28-day cycle.
  nab-paclitaxel received nab-paclitaxel intravenously at a dose of 100 mg/m2 over 30 minutes on days 1, 8, and 15 of a 28-day cycle.
  Arms: GnP

SUMMARY:
The effect of neoadjuvant chemotherapy for pancreatic cancer was gradually established. However it has been not clarified which regimen of neoadjuvant treatment for pancreatic cancer is the best.

DETAILED DESCRIPTION:
gemcitabine plus S-1 versus gemcitabine plus nab-paclitaxel

ELIGIBILITY:
Inclusion Criteria:

elective pancreatectomy for pancreatic cancer

Exclusion Criteria:

a previous cancer surgery a body weight loss of >10% during the 6 months before surgery the presence of distant metastases seriously impaired function of vital organs because of respiratory, renal, or heart disease.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
overall survival | 5 years
  postoperative survival

SECONDARY OUTCOMES:
adverse events | up to 24 weeks
  incidence of adverse events for neoadjuvant chemotherapy for pancreatic cancer

CONTACTS AND LOCATIONS:
Locations (1):
- Takehiro Okabayashi, Kochi, Japan